CLINICAL TRIAL: NCT06883604
Title: Clinical Investigation of PBS Proton Treatment in Hodgkin Lymphoma Patients - PRO-Hodgkin
Brief Title: Clinical Investigation of Proton Treatment in Hodgkin Lymphoma Patients - PRO-Hodgkin
Acronym: PRO-Hodgkin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: Sahlgrenska University Hospital (Other); University Hospital of Umeå (Unknown); Region Örebro County (Other); Karolinska University Hospital (Other); Skane University Hospital (Other); University Hospital, Linkoeping (Other); Skandion Clinic (Unknown); Swedish Cancer Society (Other)
Responsible Party: Principal Investigator, Daniel Molin, MD, PhD, associate professor, Uppsala University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-00010
Record Dates: First submitted 2025-03-08; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Hodgkin Lymphoma
Keywords: Proton therapy
MeSH Terms: conditions — Hodgkin Disease | interventions — Proton Therapy

STUDY DESIGN:
Intervention Model Description: Proton therapy, non-inferiority compared to historical cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proton therapy (Experimental): Stage 1-2A Hodgkin Lymphoma.
  Interventions: Radiation: Proton therapy.

INTERVENTIONS:
Radiation: Proton therapy. — Pencil beam scanning proton therapy to a dose of 20 or 29.75 Gy (RBE) after standard chemotherapy (2-4 ABVD).

SUMMARY:
Hodgkin Lymphoma patients with limited stage are commonly cured with limited chemotherapy followed by radiotherapy. Studies have shown a risk of late toxicity from the radiotherapy, such as second cancer, heart failure and lung toxicity. With proton therapy the dose to normal tissue can be minimised without compromising the dose to the tumor. The aim of our study is to investigate whether proton therapy can be delivered in a safe way to Hodgkin Lymphoma patients with less late side effects than conventional radiotherapy, while retaining the high cure rate.

This is a multicentre phase II study of PBS proton beam therapy in patients ≤60 years, with early stage Hodgkin Lymphoma treated with induction chemotherapy. The study is performed in a non-inferiority setting comparing with a historical population-based consecutive Swedish material. The control group was treated according to the same principles, except that the radiotherapy was delivered with photons.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of classic Hodgkin Lymphoma.
* Ann Arbour stage 1A, 1B or 2A.
* Both patients with and without risk factors, i.e. bulky disease, erythrocyte sedimentation rate (ESR)>50, more than two involved sites.
* Supra diaphragmal disease.
* Age 18-60 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2.
* Initial staging positron emission tomography/computed tomography (PET/CT).
* Induction chemotherapy including 2 cycles of ABVD for patients without risk factors and 4 cycles of ABVD for patients with risk factors.
* For patients with risk factors a CT after 2 ABVD confirming complete remission (CR) or partial remission (PR). For patients without risk factors clinical response is sufficient at inclusion, but a CT scan is recommended before start of radiotherapy.
* Radiotherapy (RT) start not later than 6 weeks after end of chemotherapy.
* Written informed consent obtained prior to any study specific procedures.
* Women of reproductive age must agree to use contraceptives during the study treatment period.

Exclusion Criteria:

* Pregnancy.
* Serious concomitant systemic disorder endangering treatment delivery.
* More than 5mm tumour motion on 4 dimensional computed tomography (4DCT) unless deep inspiration breath hold (DIBH) is used. Not applicable if target is located outside mediastinum or photon treatment is planned.
* Clinical or radiographic stable disease (SD)/ progressive disease (PD) during induction chemotherapy.
* Not able to comply with treatment and study procedures.
* No additional active malignancy except indolent lymphoma in the bone marrow, basal cell carcinoma of the skin, squamous cell carcinoma of the skin or in situ cervical cancer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2041-06 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Outcome will be measured after 1, 3, 5 and 16 years.
  Time from study entry until disease progression or death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | Outcome will be measured after 1, 3, 5 and 16 years.
  Time from diagnostic biopsy until death from any cause.
Time to progression (TTP) | Outcome will be measured after 1, 3, 5 and 16 years.
  Time from diagnostic biopsy until objective tumor progression, not includingdeath.
Absorbed dose to organs at risk. | Outcome will be measured at baseline.
  Will be collected from Dose Volume Histograms.
Patterns of failure. | Outcome will be measured after 1, 3, 5 and 16 years.
  Are failures located within or outside of the radiation field?
Acute adverse events. | Outcome will be measured within 3 months.
  The incidence of acute toxicities during treatment will be summarized by severity (based on CTCAE grades), type and relation to the study therapy. Acute adverse events are defined as occurring during or within 3 months after radiotherapy.
Long-term adverse events. | Outcome will be measured after 1, 3, 5 and 16 years.
  This study specifically includes longitudinal follow-up to assess the incidence of secondary malignant neoplasms, heart- and lung toxicity measured up to 16 years following radiotherapy. Late adverse events are defined as occurring 3 months or later.
Quality of life. | Outcome will be measured after 1, 3, 5 and 16 years.
  EORTC quality of life questionnaire (QLQ)-C30.
Quality of life. | Outcome will be measured after 1, 3, 5 and 16 years.
  EORTC quality of life questionnaire (QLQ)-Hodgkin lymphoma (HL)27.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Molin, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (6):
- Sweden (6):
  - Sahlgrenska University Hospital, Gothenburg
  - Skane University Hospital, Lund
  - Orebro University Hospital, Örebro
  - Karolinska University Hospital, Solna
  - Umea University Hospital, Umeå
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Specht L, Yahalom J, Illidge T, Berthelsen AK, Constine LS, Eich HT, Girinsky T, Hoppe RT, Mauch P, Mikhaeel NG, Ng A; ILROG. Modern radiation therapy for Hodgkin lymphoma: field and dose guidelines from the international lymphoma radiation oncology group (ILROG). Int J Radiat Oncol Biol Phys. 2014 Jul 15;89(4):854-62. doi: 10.1016/j.ijrobp.2013.05.005. Epub 2013 Jun 18. PMID 23790512
- [Background] Maraldo MV, Dabaja BS, Filippi AR, Illidge T, Tsang R, Ricardi U, Petersen PM, Schut DA, Garcia J, Headley J, Parent A, Guibord B, Ragona R, Specht L. Radiation therapy planning for early-stage Hodgkin lymphoma: experience of the International Lymphoma Radiation Oncology Group. Int J Radiat Oncol Biol Phys. 2015 May 1;92(1):144-52. doi: 10.1016/j.ijrobp.2014.12.009. Epub 2015 Feb 7. PMID 25670544
- [Background] Aznar MC, Maraldo MV, Schut DA, Lundemann M, Brodin NP, Vogelius IR, Berthelsen AK, Specht L, Petersen PM. Minimizing late effects for patients with mediastinal Hodgkin lymphoma: deep inspiration breath-hold, IMRT, or both? Int J Radiat Oncol Biol Phys. 2015 May 1;92(1):169-74. doi: 10.1016/j.ijrobp.2015.01.013. Epub 2015 Mar 5. PMID 25754634
- [Background] Petersen PM, Aznar MC, Berthelsen AK, Loft A, Schut DA, Maraldo M, Josipovic M, Klausen TL, Andersen FL, Specht L. Prospective phase II trial of image-guided radiotherapy in Hodgkin lymphoma: benefit of deep inspiration breath-hold. Acta Oncol. 2015 Jan;54(1):60-6. doi: 10.3109/0284186X.2014.932435. Epub 2014 Jul 15. PMID 25025999
- [Background] Hoppe BS, Flampouri S, Su Z, Morris CG, Latif N, Dang NH, Lynch J, Li Z, Mendenhall NP. Consolidative involved-node proton therapy for Stage IA-IIIB mediastinal Hodgkin lymphoma: preliminary dosimetric outcomes from a Phase II study. Int J Radiat Oncol Biol Phys. 2012 May 1;83(1):260-7. doi: 10.1016/j.ijrobp.2011.06.1959. Epub 2011 Oct 17. PMID 22014950
- [Background] Hoppe BS, Flampouri S, Su Z, Latif N, Dang NH, Lynch J, Joyce M, Sandler E, Li Z, Mendenhall NP. Effective dose reduction to cardiac structures using protons compared with 3DCRT and IMRT in mediastinal Hodgkin lymphoma. Int J Radiat Oncol Biol Phys. 2012 Oct 1;84(2):449-55. doi: 10.1016/j.ijrobp.2011.12.034. Epub 2012 Mar 2. PMID 22386373
- [Background] Hoppe BS, Flampouri S, Zaiden R, Slayton W, Sandler E, Ozdemir S, Dang NH, Lynch JW, Li Z, Morris CG, Mendenhall NP. Involved-node proton therapy in combined modality therapy for Hodgkin lymphoma: results of a phase 2 study. Int J Radiat Oncol Biol Phys. 2014 Aug 1;89(5):1053-1059. doi: 10.1016/j.ijrobp.2014.04.029. Epub 2014 Jun 10. PMID 24928256
- [Background] Hoppe BS, Hill-Kayser CE, Tseng YD, Flampouri S, Elmongy HM, Cahlon O, Mendenhall NP, Maity A, McGee LA, Plastaras JP. Consolidative proton therapy after chemotherapy for patients with Hodgkin lymphoma. Ann Oncol. 2017 Sep 1;28(9):2179-2184. doi: 10.1093/annonc/mdx287. PMID 28911093
- [Background] Chang JY, Li H, Zhu XR, Liao Z, Zhao L, Liu A, Li Y, Sahoo N, Poenisch F, Gomez DR, Wu R, Gillin M, Zhang X. Clinical implementation of intensity modulated proton therapy for thoracic malignancies. Int J Radiat Oncol Biol Phys. 2014 Nov 15;90(4):809-18. doi: 10.1016/j.ijrobp.2014.07.045. Epub 2014 Sep 24. PMID 25260491
- [Background] Zeng C, Plastaras JP, Tochner ZA, White BM, Hill-Kayser CE, Hahn SM, Both S. Proton pencil beam scanning for mediastinal lymphoma: the impact of interplay between target motion and beam scanning. Phys Med Biol. 2015 Apr 7;60(7):3013-29. doi: 10.1088/0031-9155/60/7/3013. Epub 2015 Mar 19. PMID 25789418
- [Background] Zeng C, Plastaras JP, James P, Tochner ZA, Hill-Kayser CE, Hahn SM, Both S. Proton pencil beam scanning for mediastinal lymphoma: treatment planning and robustness assessment. Acta Oncol. 2016 Sep-Oct;55(9-10):1132-1138. doi: 10.1080/0284186X.2016.1191665. Epub 2016 Jun 22. PMID 27332881